CLINICAL TRIAL: NCT04750694
Title: High Intensity Resistance Training Combined With Blood Flow Restricted Exercise in Elite Handball Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department of Public Health, Denmark (Other)
Responsible Party: Principal Investigator, Simon Lønbro, Teaching Associate Professor, PhD, Department of Public Health, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VEK ID 74646
Record Dates: First submitted 2020-11-17; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Hypertrophy
Keywords: The focus is blood flow restricted exercise
MeSH Terms: conditions — Hypertrophy | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT + BFRE (Experimental): High intensity Resistance training combined with Blood Flow
  Interventions: Behavioral: Resistance training
- RT (Active Comparator): Resistance training alone
  Interventions: Behavioral: Resistance training

INTERVENTIONS:
Behavioral: Resistance training — A full-training programme with high intensity followed by back squat exercise with blood flow restriction. Inflatable cuffs will be placed proximally on both thighs. The cuff pressure will be 50% of individual arterial occlusion pressure and will be maintained during the rest intervals. Participants will perform 30, 15, 15 and 15 repetitions of 30% of 1 Repetition Maximum. Totally 75 repetitions will be performed. 45 seconds rest interval between sets will be given.

SUMMARY:
Purpose of the study is: to investigate the effects of 8 weeks intervention of high intensity resistance training(HIRT) combined with Blood Flow Restricted Exercise (BFRE) compared to high intensity resistance training alone.

Detailed Description: 30 elite handball players will be randomized into 2 groups of 15 participants each. Participants will be evaluated in the week before and the week after an 8-weeks training intervention with 2 weekly sessions. Based on their baseline muscle strength the participants will be randomized into two groups: HIRT-BFRE or HIRT-HIRT. Participants in both groups will perform a full-body training programme of HIRT. After the Full-body programme, Back squat exercise with low intensity and Blood flow restriction will be performed to the HIRT-BFRE group and back squat exercise with high intensity without blood flow restriction will be performed by HIRT-HIRT. Evaluation protocol includes: muscle strength measurement with 1 repetition maximum of Back squat and knee extension, muscle mass with Dual-Energy X-ray absorptiometry, muscle thickness of the thigh with ultra sound measurement, vertical jump height with linear Encoder, sprint performance with 30m sprint time.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Ds
* Minimum of 2 years of resistance training experience
* >< Two resistance training sessions each week
* >< three handball sessions each week
* No injuries that prevent participants to perform test of maximal muscle strength
* No injuries, that affects the muscle strength or the ability to train

Exclusion Criteria:

* Elevated blood pressure (>140/90)
* Anabolic steroids or prescription-only medical products with know or potential effect on muscle hypertrophy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Maximal Muscle Strength | Baseline measurements at week 1, after four weeks of exercise at week 5 and post intervention at week 10.
  Change in 1 RM (repetition maximum) muscle strength in back squat

SECONDARY OUTCOMES:
Change in Lean body mass | Baseline measurements at week 1 and post intervention at week 10.
  Change in lean body mass assessed by Dual Energy X-ray Absorptiometry

OTHER OUTCOMES:
Jump Performance | Baseline measurements at week 1 and post intervention at week 10.
  Change in jump height. Change in vertical jump height (in cm, with Chronojump Linear Encoder Kit). Participants will perform a counter movement jump and jump as high as possible. The jump height will be recorded.
Sprint performance | Baseline measurements at week 1 and post intervention at week 10.
  Sprint performance. Change in sprint time (in seconds, with Witt speed gates). Participant will perform a 30-meter sprint on an indoor handball court. The time to perform a 30-meter sprint will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Public Health, Aarhus, Denmark